CLINICAL TRIAL: NCT06176599
Title: Clinical Study on the Treatment of Diabetic Kidney Disease With Shenxiao Yuning Decoction With Syndrome of Qi and Yin Deficiency and Blood Stasis
Acronym: SXYNT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lin Liao (Other)
Responsible Party: Sponsor-Investigator, Lin Liao, Director of Endocrinology Department, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2023(137); YXLL-KY-2023(137) (Other: The First Affiliated Hospital of Shandong First Medical University)
Record Dates: First submitted 2023-12-08; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Kidney Disease
Keywords: Shenxiao Yuning Decoction; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shenxiao Yuning decoction (Experimental): * Diabetes education
    * control of blood glucose; ③Control blood lipids；
      * Control blood pressure； ⑤Other symptomatic treatment； ⑥Shenxiao Yuning decoction：Astragalus 30g, Radix Pseudostellariae 15g, Rehmannia glutinosa 15g, Rhodiola rosea 12g，Cimicifuga 15g，Cuttlebone 15g，Poria 15g，Cicada degeneration 9g，Rheum palmatum 6g.
  Usage: Decoct by the Traditional Chinese Medicine Pharmacy of the First Affiliated Hospital of Shandong First Medical University. Put 14 doses of Chinese medicine into the decoction bag, then put it into the automatic decoction machine, add 8 L of water and soak for 30 minutes, follow the standard decoction process Decoct 28 bags of Chinese medicine liquid, each bag is 200ml. Take 200ml warmly half an hour after breakfast and dinner.
  Interventions: Drug: Shenxiao Yuning decoction; Drug: Symptomatic treatment
- Symptomatic treatment (Active Comparator): * Diabetes education: all study participants were given dietary guidance for diabetic nephropathy, low-fat, high-quality, low-protein diet, and restricted sodium intake; maintain emotional stability, quit smoking and alcohol, and exercise appropriately; ② control of blood glucose: all study participants routinely received hypoglycaemic treatment, hypoglycaemic measures are not limited (including oral hypoglycaemic drugs or insulin injection); (iii) Control of lipids: study participants with substandard lipids routinely receive lipid-lowering treatment; (iv) Control of blood pressure: those with blood pressure >140/90 mmHg should be treated with antihypertensive drugs to control blood pressure, and antihypertensive measures are not limited (CCB class, ACEI or ARB class, α, β-blockers, diuretics, etc.); ⑤ Other symptomatic treatment.
  Interventions: Drug: Symptomatic treatment

INTERVENTIONS:
Drug: Shenxiao Yuning decoction — Astragalus 30g, Radix Pseudostellariae 15g, Rehmannia glutinosa 15g, Rhodiola rosea 12g，Cimicifuga 15g，Cuttlebone 15g，Poria 15g，Cicada degeneration 9g，Rheum palmatum 6g.
  Arms: Shenxiao Yuning decoction
Drug: Symptomatic treatment — (i) Diabetes education: all study participants were given dietary guidance for diabetic nephropathy, low-fat, high-quality, low-protein diet, and restricted sodium intake; maintain emotional stability, quit smoking and alcohol, and exercise appropriately; (ii) control of blood glucose: all study participants routinely received hypoglycaemic treatment, hypoglycaemic measures are not limited (including oral hypoglycaemic drugs or insulin injection); (iii) Control of lipids: study participants with substandard lipids routinely receive lipid-lowering treatment; (iv) Control of blood pressure: those with blood pressure >140/90 mmHg should be treated with antihypertensive drugs to control blood pressure, and antihypertensive measures are not limited (CCB class, ACEI or ARB class, α, β-blockers, diuretics, etc.); ⑤ Other symptomatic treatment.

SUMMARY:
To explore the therapeutic effect of Shenxiao Yuning Decoction on albuminuria and the improvement of traditional Chinese medicine syndrome in patients with stage III diabetic kidney disease with Qi and Yin deficiency and blood stasis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for albuminuria in type 2 diabetic nephropathy, persistent albuminuria, and 2 consecutive urine microalbumin/creatinine (ACR) >30mg/g within 3 months;
* The glomerular filtration rate eGPR ≥ 60ml/min/1.73m2, and is required to remain stable during the trial (eGFR decreases ≤25% from the beginning of screening to the second week of follow-up);
* Those who are consistent with the syndrome of diabetes and kidney disease, deficiency of Qi and Yin and blood stasis;
* Gender is not limited, age is 18-75 years old, BMI≤45 kg/m2;
* Glycated hemoglobin (HbA1C) 6-11%, fasting blood glucose (FPG) ≤15 mmol/L;
* Systolic blood pressure/diastolic blood pressure (SBP/DBP) ≤180/100 mmhg (sitting);
* Those who have complete medical records, voluntarily participate in this clinical study, and sign the informed consent form.

Exclusion Criteria:

* Pregnant and lactating women;
* Acute complications of diabetes such as hypoglycemic coma, diabetic ketosis, lactic acidosis, etc. have recently occurred;
* Those combined with heart failure and myocardial infarction; combined with infections, immune diseases, and malignant tumors; combined with liver diseases (ALT, AST or ALP levels exceed three times the upper limit of normal);
* Male serum creatinine (SCr) ≥1.50 mg/d1 (114.4 μmol/L), or female serum creatinine ≥1.40 mg/dl (106.8 μmol/L);
* Those who are combined with other kidney and renovascular diseases, or those who have other causes such as excessive exercise, heart failure, febrile infections, or urinary tract infections that lead to elevated urinary microalbumin;
* Those who have used nephrotoxic drugs and antioxidants, or used systemic glucocorticoid therapy in the past 2 weeks;
* Those undergoing dialysis or kidney transplantation;
* History of bariatric surgery or other gastrointestinal surgery causing chronic malabsorption within 2 years;
* Persons with drug contraindications: pregnant or lactating women, allergic constitutions, and those allergic to the drugs used in this study;
* Those who are unable to cooperate due to severe mental illness or mental disorder;
* Those who have not signed the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Effective rate | 0 week，4 weeks
  Clinical control: Urine routine examination of urine protein qualitative turn negative, ACR normal. Apparent effect: ACR reduction ≥50%. Effective: ACR reduction ≥15%, but less than ≥50%. Ineffective No improvement in clinical manifestations and laboratory parameters.

SECONDARY OUTCOMES:
Urinary α1-MG | 0 week，4 weeks
  Charge patients for random urine measurements Urinary α1-MG
Urinary β2-MG | 0 week，4 weeks
  Collect random urine measurements from patients Urinary β2-MG
Scr | 0 week，4 weeks
  Collect the patient's fasting blood to measure Scr
BUN | 0 week，4 weeks
  Collect the patient's fasting blood to measure BUN
uric acid | 0 week，4 weeks
  Collect the patient's fasting blood to measure uric acid
Cys-C | 0 week，4 weeks
  Collect the patient's fasting blood to measure Cys-C
fasting plasma glucose | 0 week，4 weeks
  Collect the patient's fasting blood to measure fasting plasma glucose
HbA1c | 0 week，4 weeks
  Collect the patient's fasting blood to measure HbA1c
total cholesterol | 0 week，4 weeks
  Collect the patient's fasting blood to measure total cholesterol
Triglyceride | 0 week，4 weeks
  Collect the patient's fasting blood to measure Triglyceride
HDL | 0 week，4 weeks
  Collect the patient's fasting blood to measure HDL
LDL | 0 week，4 weeks
  Collect the patient's fasting blood to measure LDL
albumin | 0 week，4 weeks
  Collect the patient's fasting blood to measure albumin
Urinary microalbumin/urinary creatinine | 0 week，4 weeks
  Collect random urine samples from patients to measure urine microalbumin/urinary creatinine（mg/g）

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided